CLINICAL TRIAL: NCT06270004
Title: Effect of Nonsurgical Periodontal Therapy on Salivary Biomarkers Related to Bone Turnover in Smoker and Nonsmoker Periodontitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Aqeel Ali, Iraq ,baghdad, University of Baghdad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: nonsurgical periodontal
Record Dates: First submitted 2024-01-08; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Non Surgical Periodontal Therapy
Keywords: osteonectin; osteopontin; histatin1

STUDY DESIGN:
Intervention Model Description: smoker and non smoker patients with unstable periodontitis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nonsmoker periodontitis patients (Active Comparator)
  Interventions: Other: nonsurgical periodontal therapy
- smoker periodontitis patients (Active Comparator): cigarette smoker more the three years ago
  Interventions: Other: nonsurgical periodontal therapy

INTERVENTIONS:
Other: nonsurgical periodontal therapy — sonic scaler for scaling and polishing. Graces curettes numbers(1-2,3-4,5-6,7-8,9-10,11-12,13-14)for root surfaces debridement(RSD), instructions and motivation for dental arch

SUMMARY:
1. To assess the alteration in the level of salivary osteopontin (OPN), osteonectin(ON) and histatin-1 following NSPT in smoker and nonsmoker unstable periodontitis patients at different time intervals(one month and three months) .
2. To evaluate the response of clinical periodontal parameters ( plaque index ,bleeding on probing ,probing pocket depth ,clinical attachment loss)following NSPT in smoker and nonsmoker unstable periodontitis patients at different time intervals (one month and three months)

DETAILED DESCRIPTION:
the study include nonsurgical periodontal therapy for smoker and non smoker patients with unstable periodontitis and evaluate the clinical periodontal parameters ( plaque index, bleeding on probing , probing pocket depth ,clinical attachment loss) and assess the alteration in the level of salivary osteopontin (OPN), osteonectin(ON) and histatin-1 following NSPT in smoker and nonsmoker unstable periodontitis patients at different time intervals(one month and three months)

ELIGIBILITY:
Inclusion Criteria:

* participants will be systemically healthy without history of any systemic diseases.
* hadn't underwent periodontal treatment during the previous 6 months and not taken medication during the previous 3 months.
* present with at least 20 teeth, those who only diagnosed with 4-6 mm probing pocket depth, generalized ,unstable periodontitis who had bone loss > 30% , probing probing pocket depth at ≥4mm . Periodontitis cases were defined if clinical attachment loss was detected at ≥2 non- adjacent teeth or when buccal (facial) showed clinical attachment loss ≥3mm associated with probing pocket depth >3mm at ≥ 2 teeth .
* The patients in the smokers group will be current smokers ( cigarette smokers) with smoking habit for over 3 years

Exclusion Criteria:

* Subjects have any intraoral plaque retentive factors such as those wearing partial denture, crown and bridges, and orthodontic appliances ,furcation involved teeth, overhang filling, tooth anomaly.
* receiving antibiotic therapy during the previous 3 months.
* those with systemic diseases such as diabetes mellitus, cardiovascular or renal diseases, etc…., pregnant or lactating women, not willing to participate or continue to conduct the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of nonsurgical periodontal therapy(NSPT) on salivary biomarkers related to bone turnover in smoker and nonsmoker periodontitis patients. | baseline, one month and three months
  salivary concentration of osteopontin between smoker and nonsmoker unstable periodontitis patients following NSPT at different time intervals.

SECONDARY OUTCOMES:
Effect of nonsurgical periodontal therapy(NSPT) on salivary biomarkers related to bone turnover in smoker and nonsmoker periodontitis patients. | baseline, one month and three months
  salivary concentration of osteonectin between smoker and nonsmoker unstable periodontitis patients following NSPT at different time intervals .
Effect of nonsurgical periodontal therapy(NSPT) on salivary biomarkers related to bone turnover in smoker and nonsmoker periodontitis patients | baseline, one month and three months
  salivary concentration of histatin1 between smoker and nonsmoker unstable periodontitis patients following NSPT at different time intervals.

IPD SHARING:
Plan to Share IPD: No